CLINICAL TRIAL: NCT04477395
Title: Omega-3 Polyunsaturated Fatty Acids EPA and DHA as an Adjunct to Non-surgical Treatment of Periodontitis: a Randomized Clinical Trial
Brief Title: Omega-3 Polyunsaturated Fatty Acids in Non-surgical Treatment of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RNN/251/17/KE
Record Dates: First submitted 2020-06-22; First posted 2020-07-20 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis; Therapeutics; Fatty Acids, Unsaturated
Keywords: periodontitis; non-surgical treatment; eicosapentaenoic acid; docosahexaenoic acid
MeSH Terms: conditions — Periodontitis | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP plus fish oil (Experimental): Patients will receive scaling and root planing (SRP) supplemented with the dietary fish oil rich in omega-3 PUFAs: 2.6 g of EPA and 1.8 g DHA daily for 6 months.
  Interventions: Dietary Supplement: fish oil; Procedure: SRP only
- SRP alone (Active Comparator): Patients will receive scaling and root planing (SRP) only.
  Interventions: Procedure: SRP only

INTERVENTIONS:
Dietary Supplement: fish oil — SRP will be supplemented with the dietary fish oil rich in omega-3 PUFAs EPA and DHA for 6 months. Fish oil (BioMarine Medical, 200 ml liquid), obtained from Tasmanian deep sea shark and Norwegian cod liver and sardine, anchovy and mackerel muscle, will be administered two times a day at a dose 10 ml. Daily dose of 20 ml provides 2.6 g of EPA and 1.8 g of DHA.
  Other Names: BioMarine Medical
  Arms: SRP plus fish oil
Procedure: SRP only — Scaling and root planing will be the only method of treatment.

SUMMARY:
Periodontitis is a chronic multifactorial inflammatory disease that lead to the loss of supportive tissues around the teeth with gradual deterioration of masticatory function and esthetics, resulting eventually in the decrease of the quality of life. Host immune response triggered by bacterial biofilm is responsible for the chronic periodontal inflammation and ongoing tissue loss. Polyunsaturated fatty acids (PUFAs) omega-3 eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) have anti-inflammatory properties, thus may be used for the treatment of chronic inflammatory diseases. This study is aimed to evaluate the effect of dietary supplementation with PUFAs omega-3 in the patients with periodontitis stage III and IV.

DETAILED DESCRIPTION:
Periodontitis is highly prevalent oral disease in humans affecting nearly 50% of the population worldwide. Periodontitis is multifactorial disease individually accelerated or decelerated by different factors. One of them, a bacterial biofilm, leads to dysbiosis and raise of Gram-negative bacteria.This results in the activations of immune response and clinical signs of periodontal tissue inflammation. Host modulation therapy seems to be an adequate concept for the treatment of periodontal diseases. The main assumption of this therapy is to reduce by-stander tissue destruction, to ensure rapid resolution of inflammation or even to promote regeneration of the periodontal tissues by modifying or down-regulating the destructive aspects of the host response and by up-regulating the protective or regenerative responses The goal of the present study was to assess the effect of high-dose omega-3 PUFAs EPA and DHA on the clinical outcome of non-surgical treatment of the patients with generalized periodontitis stage III and IV. It was presumed that dietary supplementation with high-dose EPA and DHA would have the potential to induce a measurable clinical outcome as a result of reduction of inflammation and minimizing tissue damage mediated by anti-inflammatory effect of omega-3 PUFAs. To address this issue, a randomized clinical trial was designed in which EPA and DHA were supplemented in adjunction to the standard periodontal therapy, scaling and root planning (SRP). Clinical outcomes of active versus control therapies were measured in addition to the quantifications of saliva cytokines, chemokines, subgingival biofilm composition and serum levels of lipids.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 scorable teeth (not including third molars),
* ≥4 teeth with PD ≥6 mm, CAL ≥5 mm,
* radiographic evidence of bone loss more than one-third of the root length,
* no periodontal treatment performed within last 6 months.

Exclusion Criteria:

* smoking,
* diabetes,
* any diseases or disorders that compromise wound healing,
* chronic inflammatory disease, history of radio- or chemotherapy,
* nonsteroidal anti-inflammatory drug (NSAIDs) intake > 3 days,
* use of antibiotics or corticosteroids 3 months prior to the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the percent of closed pockets | 3 and 6 months
  The percent of closed pockets (PD ≤ 4 mm and BOP-) at 3 and 6 months in relation to baseline

SECONDARY OUTCOMES:
Change in the probing depth (PD) | 3 and 6 months
  Mean values of probing depth of all sites with initial PD ≥ 4 mm
Change in the clinical attachment level (CAL) | 3 and 6 months
  Mean values of clinical attachment level of all sites with initial PD ≥ 4 mm
Change in the bleeding on probing (BOP) | 3 and 6 months
  Percent of all sites with bleeding on probing
Change in the number of sites with PD ≥ 4 mm and BOP+ | 3 and 6 months
  Mean values of number of sites with PD ≥ 4 mm and BOP+

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Lewkowicz, Prof., Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Periodontology and Oral Mucosal Diseases, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stando-Retecka M, Piatek P, Namiecinska M, Bonikowski R, Lewkowicz P, Lewkowicz N. Clinical and microbiological outcomes of subgingival instrumentation supplemented with high-dose omega-3 polyunsaturated fatty acids in periodontal treatment - a randomized clinical trial. BMC Oral Health. 2023 May 13;23(1):290. doi: 10.1186/s12903-023-03018-7. PMID 37179297